CLINICAL TRIAL: NCT05689580
Title: The Influence of Ketogenic Diet on Lupus Nephritis Patients' Immunity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202001487A3C102
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-09

CONDITIONS: Systemic Lupus Erythematosus; Ketogenic Dieting
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: For Group 1, subjects will be educated by dietitian and receive two months of ketogenic diet. Then, followed by three months of washout period. Finally, they will receive dietary education and follow balanced diet for two months. For Group2, subjects will receive dietary education and follow balanced diet for two months first, then followed by three months of washout period. At last, they will receive dietary education of ketogenic diet and need to follow the ketogenic diet for two months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients received ketogenic diet then Balanced diet (Experimental): subjects will be educated by dietitian and receive two months of ketogenic diet. Then, followed by three months of washout period. Finally, they will receive dietary education and follow balanced diet for two months.
  Interventions: Dietary Supplement: Ketogenic diet; Dietary Supplement: Balanced diet
- Patients received Balanced diet then ketogenic diet (Experimental): subjects will receive dietary education and follow balanced diet for two months first, then followed by three months of washout period. At last, they will receive dietary education of ketogenic diet and need to follow the ketogenic diet for two months.
  Interventions: Dietary Supplement: Ketogenic diet; Dietary Supplement: Balanced diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — The course of the trial to medium-chain triglyceride lipid intervening 50-70% of dietary intake
Dietary Supplement: Balanced diet — Balanced diet

SUMMARY:
The study investigates the dietary habits in relation to low doses of omega-3 fatty acids in subcutaneous adipose tissue, disease activity and atherosclerosis. The low intake of omega-3 and high intake of carbohydrate among patients with SLE appear to be associated with worse disease activity, adverse serum lipids and plaque presence.Three-month-old mice received an injection of pristane or saline solution and were fed with different experimental diets: sunflower oil diet or extra virgin olive oil (EVOO) diet. After 24 weeks, mice were sacrificed, spleens were collected and kidneys were removed for immunoinflammatory detections. The study have demonstrated that EVOO diet significantly reduced renal damage and decreased cytokine: TNF-α, IL-6, IL-10 and IL-17 production.The ketogenic diet utilizes a high fat, adequate protein, low carbohydrate diet that control type of food and exchange. The aim of the present study that ketogenic diet treated in SLE patients may decrease overactive immunity and associated inflammatory markers.

DETAILED DESCRIPTION:
This study was conducted in patients with lupus nephritis at outpatient department, who are 1.more than 20 years old, 2. can accept these dietary intervention and fill out 《20200909 version4》 the consent, 3. Satisfy at least four criteria according to 1997 American College of Rheumatology Classification Criteria, 4. Under maintenance stage of disease and have more than 1gm of daily proteinuria.

These enrollees will be assigned into two groups randomly. For Group 1, subjects will be educated by dietitian and receive two months of ketogenic diet. Then, followed by three months of washout period. Finally, they will receive dietary education and follow balanced diet for two months. For Group2, subjects will receive dietary education and follow balanced diet for two months first, then followed by three months of washout period. At last, they will receive dietary education of ketogenic diet and need to follow the ketogenic diet for two months.

During the Ketogenic diet (2months) and balanced diet (2months) period, subjects were separately assessed with nutritional status evaluation and laboratory data follow-up for 4 times (Day1, 1st week, 1st month, 2nd month). During the 8 times visits , anthropometric, age, sex, height, weight, BMI, muscle girdle measurements, biochemical measurements, serum albumin, blood urea nitrogen, hemoglobin, and electrolyte, nitrogen balance, and medical records are evaluated. The course of the trial to medium-chain triglyceride lipid intervening 50-70% of dietary intake, the first day of consumption of 1/3 amount of medium chain fat, if no adverse adaptation, an increase of 1/3 volume until the full amount of intervening nutrition The division is responsible for designing menus that contain information on how to purchase special dietary formulas, calculate and cook, and possibly prepare food for future problem solving. Results were presented as mean ± SD. Statistical analysis was performed using SPSS software version 21.0. Difference in patients' dietary intake and biochemical values were compared for the significant differences at

1st, 2th month using one-way analysis of variance (ANOVA). Comparison of male and female baseline characteristics were using by unpaired t-test.

ELIGIBILITY:
Inclusion Criteria:

1. more than 20 years old
2. can accept these dietary intervention and fill out the consent
3. Satisfy at least four criteria according to 1997 American College of Rheumatology Classification Criteria
4. Under maintenance stage of disease and have more than 1gm of daily proteinuria.

Exclusion Criteria:

1. Can't cooperate the diet intervention
2. Rapid progression of renal function, or already need renal replacement therapy (Dialysis or kidney transplantation)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
urine albumin creatinine ratio | 8 times: Day1, 1st week, 1st month, 2nd month during ketogenic diet then Day1, 1st week, 1st month, 2nd month during balanced diet
  By using urine albumin creatinine ratio to determine whether the ketogenic diet could result in less proteinuria
Change in Inflammatory cytokine | 8 times: Day1, 1st week, 1st month, 2nd month during ketogenic diet then Day1, 1st week, 1st month, 2nd month during balanced diet
  By testing blood inflammatory cytokine: TNF-α, IL-6, IL-10 and IL-17 to evaluate whether the ketogenic diet could decrease systemic inflammation

SECONDARY OUTCOMES:
Change of subclass of T cells | 2 times: 2nd month during ketogenic diet then 2nd month during balanced diet
  By using flow cytometry to detect the change of subclasses of blood T cells after ketogenic diet
Change of Gut microbiota analysis | 2 times: 2nd month during ketogenic diet then 2nd month during balanced diet
  By using new generation sequencing to detect the change of gut microbiota after ketogenicdiet

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung memorial hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided